CLINICAL TRIAL: NCT03963960
Title: Evaluation of Daily Hemodialysis With Low Dialysate Flux in Unscheduled Patients With Kidney Injury Admitted to Hemodialysis
Acronym: EQUODIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical difficulties in the department due to a lack of paramedical staff and dialysis space.
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD039-19
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury; Kidney Failure, Chronic
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis with low dialysate flow (Experimental)
  Interventions: Device: Hemodialysis with low dialysate flow
- Conventional triweekly high-flow hemodialysis (Active Comparator)
  Interventions: Device: Conventional triweekly high-flow hemodialysis

INTERVENTIONS:
Device: Hemodialysis with low dialysate flow — Hemodialysis with low dialysate flow
  Arms: Hemodialysis with low dialysate flow
Device: Conventional triweekly high-flow hemodialysis — Conventional triweekly high-flow hemodialysis
  Arms: Conventional triweekly high-flow hemodialysis

SUMMARY:
The objective of the EQUODIA study is to evaluate the hemodynamic stability of hemodialysis with low dialysate flow in patients requiring emergency hemodialysis in the context of acute kidney injury or unscheduled end-stage renal disease, not in intensive care, compared to conventional triweekly high-flow hemodialysis.

Short daily hemodialysis has excellent hemodynamic tolerance, which has already been confirmed by clinical experience. This modality, commonly used in the patient's home through new machines allowing a low dialysate flow purification technique, can prove to be an innovative, effective and safe alternative for patients admitted for hemodialysis in an unscheduled situation (acute kidney injury, unscheduled end-stage renal disease not followed).

Up to now, no studies have evaluated the use of short daily hemodialysis with low dialysate flow in patients with acute kidney injury or unscheduled end-stage renal disease, requiring the initiation of emergency extra-renal purification.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 years of age or older
* Patient requiring unscheduled hemodialysis for end-stage renal disease or acute kidney injury
* Patient able to understand the protocol
* Patient who has agreed to participate in the study and has given express oral consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient with more than one dialysis session
* Intensive care patient (need for vasoactive amine infusion, non-invasive ventilation, assisted ventilation)
* Patient participating in interventional clinical research involving a drug/medical device
* Patient under guardianship, curator, deprived of liberty
* Pregnant or breastfeeding patient, or with the ability to procreate without effective contraception
* Patient refusing to participate
* Patient unable to understand the protocol and/or give express oral consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of hypotension episodes | During the first two weeks of dialysis
  Decrease of ≥ 20 mmHg systolic blood pressure in regard to pre-dialysis value, associated with symptoms such as abdominal pain, yawn, nausea, vomiting, cramps, anxiety, dizziness, malaise and/or loss of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Natalia TARGET, PH, Study Director — CHD Vendée de la Roche sur Yon
Locations (1):
- Centre Hospitalier Départemental Vendée, La Roche-sur-Yon, France